CLINICAL TRIAL: NCT06428149
Title: Wound Healing After Different Types of Papilla Incision in Periodontal Reconstruction Surgery. a Randomized Clinical Trial
Brief Title: Three Types of Papilla Incision in Periodontal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2937/2020
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Midline interproximal soft-tissue incision (Experimental): Marginal approach by midline interproximal soft tissue incision and a limited papilla elevation to the buccal aspect will be made for treating isolated periodontal defect. Enamel matrix derivates will be applied on the debrided root surfaces.
  Interventions: Procedure: Midline interproximal soft-tissue incision
- Marginal approach by palatal incision (Active Comparator): A small incision in the palatal aspect and a limited papilla elevation to the buccal aspect will be made for treating isolated periodontal defect. Enamel matrix derivates will be applied on the debrided root surfaces.
  Interventions: Procedure: Marginal approach by palatal incision
- Minimally invasive surgical technique (Active Comparator): The incision of the defect-associated papilla will be performed according to the principles of the papilla preservation techniques. Enamel matrix derivates will be applied on the debrided root surfaces. Stable primary closure of the flaps will be obtained with internal modified mattress sutures.
  Interventions: Procedure: Minimally invasive surgical technique

INTERVENTIONS:
Procedure: Midline interproximal soft-tissue incision — Firstly, the marginal tissue will be elevated around the periodontal defect, through the tunneling of the tissues, entering through the gingival sulcus and the periodontal pocket of the teeth involved in the defect periodontal. Once the marginal tissues have been disinserted to full thickness, the soft supra-alveolar component of the defect to be reconstructed will be stretched, in a buccal direction, with a blunt instrument, applying pressure on the lingual aspect. Visualizing the midpoint of the interproximal tissue, the papilla will be dissected at its midpoint, entering through the mesial aspect, with the scalpel blade perpendicular to the central axis of the teeth.
  Arms: Midline interproximal soft-tissue incision
Procedure: Marginal approach by palatal incision — First, an incision will be made in the palatal aspect of the interproximal papilla, at the base of the papilla, parallel to the axis of the tooth until touching the palatine alveolar crest, in order to detach and move the papilla from its base, attached to the vestibular flap. From the palatal incision the interproximal tissue will be elevated towards the buccal until the buccal bone crest is exposed.
  Arms: Marginal approach by palatal incision
Procedure: Minimally invasive surgical technique — The defect will be accessed through an incision at the base of the papilla on the vestibular aspect. Depending on the anatomy of the interproximal space, two types of incisions will be made: simplified papilla preservation flap (SPPF) when the width of the interproximal space is equal to or less than 2 mm, or modified papilla preservation technique (MPPT) when the width is greater than 2 millimeters. The interproximal incision will extend intrasulcular on the lingual and buccal aspect of the teeth adjacent to the defect, and mesio-distally it will extend as necessary to allow access to the defect and its debridement. The papilla will move from its base towards the palatine.
  Arms: Minimally invasive surgical technique

SUMMARY:
Three types of papilla incision in periodontal reconstruction techniques will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontal disease.
* Active residual pockets associated with intraosseous defects that did not resolve with non-surgical treatment after 1 year of maintenance.
* Intraosseous lesions with probing depth greater than 5 mm or extension of the radiographic defect greater than 4 mm.
* Plaque index and bleeding index less than 30%.

Exclusion Criteria:

* Systemic disease that contraindicates periodontal surgery.
* Pregnant women.
* Third molars or teeth with incorrect endodontic or restorative treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing | 12 months
  Bleeding on probing could be positive or negative
Clinical attachment level (CAL) | 12 months
  Clinical attachment level will be assessed with a periodontal probe, measured in mm from the cementoenamel junction (CEJ) to the bottom of the pocket
Probing pocket depth (PD) | 12 months
  Probing pocket depth will be assessed with a periodontal probe, measured in mm from the gingival margin to the bottom of the pocket
Recession (REC) | 12 months
  Recession, will be assessed with a periodontal probe, measured in mmm on the buccal aspect, from the CEJ to the gingival margin zenith.
Location of the tip of the papillae (TP) | 12 months
  Location of the tip of the papillae. Taking as reference the level of the mid-axis of the tooth, will be measured the distance from the CEJ at the zenith of the tooth to the tip of the papilla. A positive value will be recorded when the tip of the papillae is located coronally to the CEJ and a negative value otherwise. This outcome will be assessed with a periodontal probe and measured in mm.
Keratinized tissue width (KT) | 12 months
  Keratinized tissue width will be assessed with a periodontal probe, measured in mm on the buccal aspect, from the gingival margin to the mucogingival line.

SECONDARY OUTCOMES:
Supra-alveolar attachment gain (SUPRA-AG) | 12 months
  Subtracting the 12 month CAL from the intrasurgically Bone Component-CEJ will provide the SUPRA-AG result.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Murcia, Spain